CLINICAL TRIAL: NCT00194883
Title: Cytokines and Growth in Children With CRI and ESRD
Brief Title: Effect of Cytokines on Growth of Children With Chronic Kidney Failure
Status: Suspended | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0596-363
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Chronic Renal Insufficiency
Keywords: Recombinant Human Growth Hormone; Leptin; Cytokines; Chronic Renal Insufficiency; Children
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Growth Hormone

INTERVENTIONS:
Drug: Recombinant Human Growth Hormone

SUMMARY:
Children with chronic kidney failure often do not grow well. This study examines the possible causes of growth failure in these children and the response to recombinant human growth hormone. The growth hormone-insulin-like growth factor axis will be studied in relation to biochemical and immunological parameters as well as body compositional changes pre- and post recombinant human growth hormone therapy.

DETAILED DESCRIPTION:
Children with chronic renal failure (CRF; estimated creatinine clearance less than 75ml/min/1.73 m2) and end-stage renal disease (ESRD; dialysis dependent) have marked growth retardation and often do not achieve their expected height based on genetic potential despite adequate caloric supplementation, and more recently, rhGH treatment. Resistance to both endogenous and rhGH has been proposed to account for much of this growth failure, although the specific mechanisms remain unknown. Possibilities include insensitivity to GH and an inappropriate production of IGF-I and/or a reduced bioavailability secondary to an altered GH-IGF axis. Abnormalities in the GH/IGF-I axis may result in an inability of the growth plate chondrocyte to respond appropriately. Studies combining data on nutritional parameters, changes in body composition and bone density, bone turnover and the GH-IGF axis-related proteins in children with CRF and ESRD are lacking. We propose to further characterize the specific mechanisms underlying impaired growth in pre-pubertal and pubertal children with CRF or ESRD and growth failure prior to and after the initiation of rhGH therapy. The Specific Aims of this proposal are designed to allow a more efficacious use of rhGH in maximizing growth in these children. In this study measurements of total body composition, i.e., lean body mass, fat mass and bone mineral content will be made using dual photon X-ray absorptiometry. Bone mineral density will also be determined. These studies will be correlated with anthropometric, biochemical and nutritional assessments of patients before and during rhGH treatment. Letin and cytokines will be concomitantly measured. Bone collagen turnover will be quantitated using pyridinoline and deoxypyridinoline cross-links excretion (in CRF patients) and serum levels of collagen type I C-terminal propeptide (CICP) concomitant with the above measurements. Bone turnover will be further assessed by looking at additional biochemical markers of bone metabolism such as osteocalcin and bone alkaline phosphatase. Serum levels of IGF-I, IGF-II, intact and fragmented IGFBP-1, -2,-3, and GH and GH-binding activity will be determined before and during rhGH therapy and correlated to measurements made in the other studies. These studies will help elucidate the differences in rhGH responsiveness in this population. Taken together, the above studies will substantially advance our understanding of how rhGH improves growth in children with CRF and ESRD.

ELIGIBILITY:
Inclusion Criteria:

* Current height < 2SD (or < 3rd percentile) for chronological age
* Chronic renal failure (estimated creatinine clearance <75 mL/min/1.73m2) or ESRD (as defined by receiving maintenance HD or PD)
* Age < 21 years and /or growth potential demonstrable by bone age

Exclusion Criteria:

* Unable or unwilling to adhere to the protocol
* Additional diagnoses that could impair responsiveness to GH, e.g. dwarfism syndromes, significant extra-renal organ disease, e.g. chronic liver disease, or chronic corticosteroid therapy

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 1997-04; Study Completion 2003-05

PRIMARY OUTCOMES:
To examine the efficacy of recombinant human growth hormone in improving growth velocity in prepubertal children with growth failure secondary to chronic kidney disease.

SECONDARY OUTCOMES:
To examine how recombinant human growth hormone effects body composition, the GH-IGF axis proteins and biochemical/immunological parameters in children with growth failure secondary to chronic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: Valerie L Johnson, M.D., Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States